CLINICAL TRIAL: NCT00924911
Title: A Two Part Single Dose, Randomized, Balanced, Crossover Study to Assess the Relative Bioavailability of Three Formulations, Drug Interaction and Food Effect on an GSK1322322 in Healthy Subjects
Brief Title: Relative Bioavailability Study in Healthy Subjects
Acronym: PDF112034
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 112034
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Infections, Bacterial
Keywords: GSK1322322, relative bioavailability, single dose, food effect, H2 blocker, healthy subjects, open label, PIB, tablet
MeSH Terms: conditions — Bacterial Infections | interventions — GSK1322322

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): A 4 way crossover of three GSK1322322 tablet formulations and GSK1322322 powder in bottle
  Interventions: Drug: GSK1322322
- Part 2 (Experimental): A 3 way crossover of a GSK1322322 tablet with a high fat meal, with Ranitidine, and with Ranitidine and Vitamin C.
  Interventions: Drug: GSK1322322

INTERVENTIONS:
Drug: GSK1322322 — Four different formulations of 1000mg of GSK1322322
  Arms: Part 1
Drug: GSK1322322 — GSK1322322 1000mg
  Arms: Part 2

SUMMARY:
Part 1 of this study will assess the relative bioavailability of GSK1322322 administered as one of three investigational tablets compared to powder in a bottle formulation. Pharmacokinetics of these three tablets will be evaluated and the investigation tablet with the optimal PK profile will be progressed to Part 2. In Part 2 the investigational tablet selected from Part 1 will be coadministered with food alone, an H2 blocker alone, or an H2 blocker given in combination with ascorbic acid to evaluate the effect on GSK1322322 pharmacokinetics. Plasma GSK1322322 PK profile, safety, and tolerability will be assessed from each dose group.

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female is eligible to enter and participate in this study if she is of Non-childbearing potential
* Male subjects must agree to use one of the contraception methods listed in the protocol Body weight greater than or equal to 50 kg and body mass index between 18.5-29.9 kg/m2 inclusive.

Capable of giving written informed consent

* QTcB less than 450 msec; or QTc less than 480 msec in subjects with Bundle Branch Block on Screening ECG.
* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%)

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined in the protocol.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive human chorionic gonadotropin test at screening or prior to dosing.
* Lactating females.
* Subjects who have asthma or a history of asthma within the past 6 months.
* History of smoking or history of regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, satsuma, ugli, tangerine, and tangelo, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04-27 (Actual); Primary Completion 2009-07-09 (Actual); Study Completion 2009-07-09 (Actual)

PRIMARY OUTCOMES:
GSK1322322 Blood PK as described in the protocol | 48 hours

SECONDARY OUTCOMES:
Safety parameters including adverse events, clinical laboratory tests, concomitant medications, electrocardiograms, and vital signs. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Naderer OJ, Dumont E, Zhu J, Kurtinecz M, Jones LS. Effect of H2 blockade and food on single-dose pharmacokinetics of GSK1322322, a peptide deformylase inhibitor antibacterial. Antimicrob Agents Chemother. 2013 Jun;57(6):2556-61. doi: 10.1128/AAC.02505-12. Epub 2013 Mar 25. PMID 23529727
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 112034 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112034?search=study&study_ids=112034#rs
- Available data/document: Informed Consent Form: 112034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register